CLINICAL TRIAL: NCT06035588
Title: Efficacy in the Reduction of Hypersensitivity During Home Whitening With 16% Carbamide Peroxide Applied on Alternate Days: a Randomized Clinical Trial
Brief Title: Effectiveness of 16% Carbamide Peroxide in Reducing Hypersensitivity During Alternate-day Home Bleaching
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Rey Juan Carlos (Other)
Responsible Party: Principal Investigator, Isabel Giráldez de Luis, Lecturer of Department for Conservative Dentistry at Rey Juan Carlos University, Universidad Rey Juan Carlos
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: URJC University
Record Dates: First submitted 2023-09-06; First posted 2023-09-13 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Dental Hypersensitivity; Teeth Whitening
Keywords: bleaching; hipersensitivity; whitening; at-home; carbamide

STUDY DESIGN:
Intervention Model Description: Each volunteer will be given 3 syringes of 16% carbamide peroxide bleaching gel to use on the splint. Volunteers will be instructed to use the whitening gel once a day for 2 hours, completing a total of 3 weeks of whitening procedure. Depending on the randomization, the whitening procedure will be performed on alternate days or daily. In the upper arch, the teeth to be whitened will be from 15 to 25 and in the lower one from 35 to 45.
Who Masked: Investigator, Outcomes Assessor
Masking Description: The present study presents blinding of both the evaluator and the person who will carry out the statistical analysis, and therefore double-blind. The evaluators are considered blind in this study because they do not know the randomization of the patients, being a blind study. The operator and patients know the groups in which they are assigned, due to the delivery and placement of the splints.
  A block randomization of the treatment applied to the patients will be carried out, to ensure that the sample size is similar in both groups. The operator will open an envelope for the group's allocation. The assignment of the groups will be carried out using opaque, sealed and sequentially numbered envelopes. The operator will open the envelope when the splints are delivered, and will give the pertinent explanations to the patient. Data will be collected from each patient that may influence treatment results such as age, sex, initial color, systemic pathologies and pharmacological treatments.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Daily whitening (Active Comparator): Volunteers should whiten daily with a whitening tray from 15 to 25 and 35 to 45 for 2 hours. This procedure will last 3 weeks.
  Interventions: Other: Daily whitening
- Alternate whitening (Experimental): Volunteers will bleach for 3 weeks with 16% carbamide peroxide, alternating one rest day for each placement day. They will wear a whitening tray from 15 to 25 and from 35 to 45 for 2 hours.
  Interventions: Other: Alternate whitening

INTERVENTIONS:
Other: Daily whitening — Daily application of a 16% carbamide peroxide bleaching gel in volunteers without sensitivity.
  Arms: Daily whitening
Other: Alternate whitening — Volunteers will apply the whitening gel at 16% carbamide peroxide, alternating a rest day with an application day. Patients should not be sensitive before starting the study.
  Arms: Alternate whitening

SUMMARY:
The concentration of 16% carbamide peroxide is the highest concentration that European regulations allow for use in home whitening (Council directive 2011/84/EU). This concentration allows for faster results, but instead patients may suffer more frequently from dental sensitivity. The most commonly described side effect of all whitening procedures is the appearance of dentin hypersensitivity, hence the efforts to counteract or overcome this adverse effect.

The objective of the study is to clinically evaluate the difference in dental hypersensitivity produced by home dental whitening treatment using 16% carbamide peroxide in a tray for two hours daily applied daily or every other day for three weeks.

DETAILED DESCRIPTION:
Volunteers will be instructed to use the whitening gel once a day for 2 hours, completing a total of 3 weeks of whitening procedure. Depending on the randomization, the bleaching procedure will be performed every other day or daily. In the upper arch, the teeth to be whitened will be from 15 to 25. The evaluations of efficacy, dental sensitivity and satisfaction will be carried out in the upper and lower arch. The color will be recorded before, weekly for 1 month, 6 months and 12 months after finishing the treatment. Shade assessment using the subjective method will be recorded with the Vita Classical color scale (Vita Zahnfabrik, Bad Säckingen, Germany), it will also be determined with the Vita 3D-MASTER scale (Vita Zahnfabrik, Bad Säckingen, Germany). For objective evaluation, the Vita Easyshade spectrophotometer (Vita Zahnfabrik, Bad Säckingen, Germany) will be used, according to the CIEL*a*b* system.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18 years.
* Patients with vital teeth without restorations, single crowns, implants and/or bridges at the level of the anterior teeth.
* Absence of cavities in the teeth to be whitened.
* Patients with satisfactory oral hygiene and periodontally healthy, who are not undergoing periodontal maintenance and who do not use chlorhexidine mouthwashes. Patients with recessions without presenting sensitivity will be included.
* Absence of sensitivity, measured with the application of air with the dental team's syringe.
* Patients whose canines have at least an A2-A3 shade (VITA Classic® Guide).

Exclusion Criteria:

* Patients who have previously undergone whitening (less than 5 years).
* Patients undergoing orthodontic treatment.
* Patients with white spots or alterations in the development of enamel or with stains.
* Patients with a history of trauma to anterior teeth.
* Patients who require internal whitening.
* Smokers.
* Pregnant or lactating.
* Patients with allergies to any whitening component.
* Patients presenting alterations of the oral mucosa (desquamative gingivitis, oral lichen planus, leukoplakia, etc.).
* Patients with medical conditions considered by the researchers that may compromise the study or the individual safety of the patient.
* Patients with poor oral hygiene.
* Patients with previous hypersensitivity.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2024-01-06 (Actual); Primary Completion 2025-02-27 (Actual); Study Completion 2025-09-01 (Actual)

PRIMARY OUTCOMES:
Dental Sensitivity Visual Analog Scale (VAS) 0-10 | 3 weeks
  The aim of this study is to clinically evaluate the incidence of tooth sensitivity induced by home whitening with 16% carbamide peroxide applied in a tray for two hours daily or every other day for three weeks. For the assessment, the operators will apply air to the cervical area of the upper and lower canines and ask the patient if he/she experienced sensitivity at any time during the treatment.

SECONDARY OUTCOMES:
Whitening Efficacy CIEL*a*b* | 1 month
  To assess whether the efficacy of the 16% carbamide peroxide bleaching treatment described above when used every other day is the same as when used every day, or whether there is a difference in bleaching efficacy. This will be determined at check-ups by measuring the upper and lower canines with the Vita EasyShade V® spectrophotometer, based on the CIEL*a*b* system, according to the CIELAB system, CIEDE2000 and the whiteness index. Where L* represents the value from 0 (black) to 100 (white) and a* and b* represent the colour, where a* is the measurement along the red-green axis and b* is the measurement along the yellow-blue axis. In addition, the operators will take shade readings on all 4 canines using the VITA Classical and 3D-MASTER guides.

OTHER OUTCOMES:
Gingival irritation VAS (0-10) | 3 weeks
  Using the Visual Analogue Scale, compare the presence of gingival irritation after every other day bleaching with 16% carbamide peroxide compared to daily application. The patient should rate the gingival irritation experienced on a scale of 0 to 10, with 10 being very irritating and 0 being not irritating at all.
Patient's oral quality of life (OHIP-14) | 1 month
  The impact of treatment outcome on the patient's oral quality of life (OHIP-14) will be assessed using a questionnaire after 16% carbamide peroxide home bleaching. The patient will complete a 14-question questionnaire on a daily basis, regardless of which group he/she belongs to, daily or alternate application.

CONTACTS AND LOCATIONS:
Locations (1):
- Isabel Giraldez de Luis, Alcorcón, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No
The results obtained will only be shared once they have been published in an impact journal.

REFERENCES:
- [Background] Cardoso PC, Reis A, Loguercio A, Vieira LC, Baratieri LN. Clinical effectiveness and tooth sensitivity associated with different bleaching times for a 10 percent carbamide peroxide gel. J Am Dent Assoc. 2010 Oct;141(10):1213-20. doi: 10.14219/jada.archive.2010.0048. PMID 20884923
- [Background] Chagas AS, Freitas KMS, Cancado RH, Valarelli FP, Canuto LFG, Oliveira RCG, Oliveira RCG. Level of satisfaction in the use of the wraparound Hawley and thermoplastic maxillary retainers. Angle Orthod. 2020 Jan;90(1):63-68. doi: 10.2319/031319-197.1. Epub 2019 Jul 22. PMID 31335161
- [Background] de Geus JL, Wambier LM, Boing TF, Loguercio AD, Reis A. At-home Bleaching With 10% vs More Concentrated Carbamide Peroxide Gels: A Systematic Review and Meta-analysis. Oper Dent. 2018 Jul/Aug;43(4):E210-E222. doi: 10.2341/17-222-L. PMID 29949477